CLINICAL TRIAL: NCT00494182
Title: A Phase II Study of Sorafenib in Combination With Carboplatin and Paclitaxel in Metastatic or Recurrent Head and Neck Squamous Cell Cancer
Brief Title: Sorafenib in Combination With Carboplatin and Paclitaxel in Treating Participants With Metastatic or Recurrent Head and Neck Squamous Cell Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0940; NCI-2018-01836 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2006-0940 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Squamous Cell Carcinoma of the Hypopharynx; Metastatic Squamous Cell Carcinoma of the Larynx; Metastatic Squamous Cell Carcinoma of the Oral Cavity; Metastatic Squamous Cell Carcinoma of the Oropharynx; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Carboplatin; Paclitaxel; Taxes; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (carboplatin, paclitaxel, sorafenib) (Experimental): Participants receive carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1, and sorafenib PO BID on days 2-19. Treatment repeats every 21 days for up to 6 courses. Starting with course 7, participants receive sorafenib PO daily in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Sorafenib

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Sorafenib — Given PO
  Other Names: BAY 43-9006

SUMMARY:
This phase II trial studies how well sorafenib works with carboplatin and paclitaxel in treating participants with head and neck squamous cell cancer that has spread to other parts of the body or that has come back. Drugs used in chemotherapy, such as sorafenib, carboplatin, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the progression free survival of the combination of sorafenib (BAY 43-9006), carboplatin, and paclitaxel in patients with recurrent or metastatic squamous cell cancer of the head and neck (SCCHN).

SECONDARY OBJECTIVES:

I. Response rate, toxicity, safety profile, exploratory biomarker data, and overall survival.

OUTLINE:

Participants receive carboplatin intravenously (IV) over 30 minutes and paclitaxel IV over 3 hours on day 1, and sorafenib orally (PO) twice daily (BID) on days 2-19. Treatment repeats every 21 days for up to 6 courses. Starting with course 7, participants receive sorafenib PO daily in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up between 21-35 days.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
* Patients must have cytologically or histologically proven recurrent or metastatic squamous cell cancer of the head and neck (SCCHN) from the primary tumor or lymph nodes of the oral cavity, larynx, oropharynx, or hypopharynx.
* No prior systemic chemotherapy for patients who present with metastatic disease. For patients with recurrent head and neck squamous cell carcinoma, prior chemotherapy is allowed if it was given as part of their definitive therapy. If patients have received prior combined modality therapy, they must be off therapy for at least 6 months.
* Patients must have at least 1 evaluable lesion. Lesions must be evaluated by computed Tomography (CT) scan or magnetic resonance imaging (MRI).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-1.
* Controlled blood pressure (defined as systolic blood pressure [BP] =< 140 mmHg and diastolic =< 85 mmHg).
* Hemoglobin >= 9.0 g/dL within 7 days prior to start of first dose.
* Absolute neutrophil count (ANC) >= 1,500/mm^3 within 7 days prior to start of first dose.
* Platelet count >= 100,000/mm^3 within 7 days prior to start of first dose.
* Total bilirubin =< 1.5 times the upper limit of normal (ULN) within 7 days prior to start of first dose.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (=< 5 x ULN for patients [pts] with [w/] liver involvement) within 7 days prior to start of first dose.
* International normalized ratio (INR) =< 1.5 and partial thromboplastin time (PTT) within (w/in) normal limits within 7 days prior to start of first dose.
* Serum creatinine =< 1.5 ULN or creatinine clearance (CrCl) >= 45 mL/min for patients (pts) w/ creatinine levels above institutional normal within 7 days prior to start of first dose.
* Amylase & lipase < 1.5 x the ULN within 7 days prior to start of first dose.
* Urinalysis (UA) must show less than 1+ protein in urine, or the pt will require a repeat UA. If repeat UA shows 1+ protein or more, a 24 hour urine collection will be required & must show total protein =< 1000 mg/24 hour to be eligible.
* Women of childbearing potential (not surgically sterilized or at least 2 years postmenopausal) must have a negative serum or urine pregnancy test performed within 7 days prior to the start of treatment.
* Women of childbearing potential and men must agree to use adequate contraception (abstinence; hormonal or barrier method of birth control) prior to study entry, for the duration of study participation and 3 months after end of treatment. Should a woman become pregnant while participating or the partner of a patient participating in this study becomes pregnant, they should inform their treating physician immediately.

Exclusion Criteria:

* Congestive heart failure (CHF) > class II New York Heart Association (NYHA); active coronary artery disease (myocardial infarction [MI] more than 6 months prior to study entry is allowed); or serious cardiac ventricular arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
* Uncontrolled hypertension defined as systolic blood pressure > 140 mmHg or diastolic pressure > 85 mmHg despite optimal medical management.
* Known history of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C.
* Active clinically serious infections (i.e. patients currently taking antibiotics) (grade 2 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events (CTCAE) version 3.0).
* Evidence or history of central nervous system (CNS) disease, including primary brain tumors, seizures disorders, or any brain metastasis.
* Thrombotic or embolic events such as cerebrovascular accident, deep vein thrombosis or pulmonary embolism. History of transient ischemic attack is allowed.
* Evidence or history of bleeding diathesis or coagulopathy.
* History of/or current evidence of hemoptysis (bright red blood of ½ teaspoon or more).
* Peripheral neuropathy >= grade 2 (NCI-CTC version 3.0).
* Anticancer chemotherapy or immunotherapy: anticancer therapy is defined as any agent or combination of agents with clinically proven anticancer activity administered by any route with the purpose of affecting the cancer, either directly or indirectly, including palliative and therapeutic endpoints.
* Radiotherapy to the target lesions within 3 weeks of start of first dose. Toxicities from radiotherapy must have resolved prior to start of first dose.
* No major surgery, open biopsy or significant traumatic injury within 4 weeks of start of first dose.
* Serious, non-healing wound, ulcer, or bone fracture.
* Granulocyte growth factors (G-CSF), within 3 weeks of study entry.
* Patients taking chronic erythropoietin are permitted provided no dose adjustment is made within 2 months prior to start of first dose.
* Pregnant or breastfeeding patients.
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Known or suspected allergy to any recombinant human antibodies, or compounds of similar chemical or biologic composition to sorafenib or any of the drugs in this study.
* Any condition that is unstable or could jeopardize the safety or compliance of the patient in the study.
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in the study EXCEPT cervical cancer in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis and T1) or any cancer curatively treated > 3 years prior to study entry.
* Known or suspected allergy to sorafenib (BAY 43-9006) or any agent given in association with this trial.
* Any malabsorption conditions.
* Therapeutic anticoagulation with warfarin, heparins, or heparinoids.
* Patients taking phenytoin, carbamazepine, and phenobarbital.
* Patients taking rifampin and/or St. John's Wort.
* Patients who are candidates for curative surgery or radiotherapy.
* The patient has progressed within 6 months after completion of curative intent (definitive) treatment for localized/locoregionally advanced disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-04-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective overall response rate | Up to 12 years
  The rate of response to the treatment will be estimated, and the 95% confidence interval will be calculated.
Time to progression | Up to 12 years
  Kaplan-Meier estimates of time to progression will be provided. Time to progression will be calculated from the first date of receiving study drug until documented progressive disease. Participants without tumor progression at the time of analysis will be censored at the date of their last tumor assessment. Log-rank test will be applied to test the differences in survivals between levels of prognostic factors.
Progression-free survival | Up to 12 years
  Kaplan-Meier estimates of progression-free survival will be provided. Progression-free survival will be calculated from the first day of receiving study drug until documented progressive disease or death due to any cause (if death occurs before progression). Log-rank test will be applied to test the differences in survivals between levels of prognostic factors.
Biomarkers | Up to 12 years
  The following biomarkers may be measured where appropriate, dependent on sample availability: phosphorylated ERK, phosphorylated VEFGR-2, p53 expression, CD31, CD34 and CD105 expression, HIF-1 alpha, HIF-2 alpha, Glut-1, CAIX, VHL and p53 mutational status, methylation status, blood cell RNA expression profiling, protein pattern profiling, Her-2, VEGF, and VEFGR2 expression. Correlation with clinical outcomes will be attempted. The association among various continuous and discrete variables will be assessed first by the exploratory data analysis using scatter plot matrix, box plots, BLiP plot. Correlation among continuous variables will be examined by Pearson or Spearman rank correlation coefficients. The association between discrete variables will be tested by Chi-square or Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: George Blumenschein, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org